CLINICAL TRIAL: NCT05790993
Title: Clinical Evaluation of the Bioli IOL Delivery System (BIOLI-D)
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOLI012021
Record Dates: First submitted 2023-02-13; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Cataract surgery is one of the most frequent surgeries carried out in the world. After cataract extraction an intraocular lens (IOL) is implanted in order to compensate for the crystalline lens power and correct patient's vision. In order to allow cataract extraction and IOL insertion, during the surgery a small incision is performed by the surgeon. This incision is performed using surgical knives, and a smaller incisión is associated with less postoperatory inflammation, faster corneal wound healing, and faster visual recovery. Several studies reported the importance of smaller incisions to reduce the risk of surgically induced astigmatism.

In order to implant the IOL through this small incision, the IOL must be preloaded in a injector that allows introducing the IOL eficiently and consistently. The manual injector BIOLI manufactured by AST Products (model D), CE approved, is designed specifically to allow the IOL insertion safely, precisely, and controllably. Among the main characteristics of this delivery system is its design to minimize the incision size widening while inserting the IOL.

The present retrospective study aims to provide more information with regards to the clinical efficacy of the BIOLI-D delivery system for the implantation of the trifocal Asqelio TFLIO130C IOL in patients submitted to cataract surgery. This will be assessed by analyzing the change in incision size after IOL implantation and the incidence of adverse events during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years or older submitted to cataract surgery and implanted with Asqelio trifocal TFLIO130C IOL using the BIOLI-D delivery system.
* Patients submitted to bilateral cataract surgery.
* Transparent ocular media, other than the bilateral cataract.

Exclusion Criteria:

* Preoperatory corneal astigmatism greater than 0.75D
* Corneal surgery or trauma prior to cataract surgery Irregular cornea
* Choroidal hemorrhage
* Microftalmos Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Concomitant ocular disease
* Not age-related cataract
* Severe optic nerve atrophy
* Diabetic retinopathy
* Proliferative diabetic retinopathy
* Amblyopia
* Extremelly shallow anterior chamber
* Severe chronic uveitis
* Rubella
* Mature/dense cataract difficulting fundas assessment preoperatively
* Prior retinal detachment
* Concurrent participation in another investigation with medication or clinical devices

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bilateral cataract submitted to cataract surgery by phacoemulsification and implantation of Asqelio trifocal TFLIO130C IOL using the BIOLI-D delivery system
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Incision size after incision | Immediately after clear incision is performed
  Determined using a Capsulorhexis Incision Gauge Set, in mm.
Incision size before IOL implantation | Immediately after phacoemulsification is complete
  Determined using a Capsulorhexis Incision Gauge Set, in mm.
Incision size after IOL implantation | Immediately after IOL implantation
  Determined using a Capsulorhexis Incision Gauge Set, in mm.
Adverse events | During or after the surgical procedure
  Incidence of adverse events related to the use of the device, coded according to the Medical Dictionary for Regulatory Activities, and analyzed per eye (ocular), and per subject (non ocular)

SECONDARY OUTCOMES:
Best corrected visual acuity | Before surgery
  Visual acuity in LogMAR units with best correction for distance, evaluated at a distance of 4m using ETDRS optotype
Best corrected visual acuity | One month after surgery
  Visual acuity in LogMAR units with best correction for distance, evaluated at a distance of 4m using ETDRS optotype
Refractive error PreOp | Before surgery
  Manifest refraction before surgery in Diopters
Refractive error PostOp | One month after surgery
  Manifest refraction after surgery in Diopters
Intraocular Pressure (IOP) | Before surgery
  Preoperative intraocular pressure measured in mmHg
Cataract grading | Before surgery
  Cataract grading before surgery using the LOCS III grading system

CONTACTS AND LOCATIONS:
Locations (1):
- OftalVist Alicante, Alicante, Spain